CLINICAL TRIAL: NCT06977061
Title: A Single-Arm, Open-Label Phase II Clinical Study of Fruquintinib Combined With Sintilimab and Stereotactic Body Radiation Therapy (SBRT) for the Second-Line and Higher-Line Treatment of Gastric or Gastroesophageal Junction Adenocarcinoma With Oligometastatic Progression
Brief Title: Efficacy and Safety of Fruquintinib Combined With Sintilimab and Stereotactic Body Radiation Therapy (SBRT) for the Second-line and Higher-line Treatment of Gastric or Gastroesophageal Junction Adenocarcinoma With Oligometastatic Progression
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Queling Liu (Other)
Responsible Party: Sponsor-Investigator, Queling Liu, Deputy Chief Physician, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IITI2024099
Record Dates: First submitted 2025-04-30; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Gastric Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fruquintinib Combined with Sintilimab and Stereotactic Body Radiation Therapy (Experimental)
  Interventions: Drug: Fruquintinib Combined with Sintilimab and Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Fruquintinib Combined with Sintilimab and Stereotactic Body Radiation Therapy — no other intervention

SUMMARY:
Efficacy and safety of fruquintinib in combination with sintilizumab and SBRT in the treatment of oligonadenocarcinoma progression in the stomach or gastroesophageal junction

DETAILED DESCRIPTION:
To explore the efficacy and safety of the combination of fruquintinib, sintilimab and SBRT for the treatment of gastric or gastroesophageal junction adenocarcinoma with oligometastatic progression in the second-line and higher-line settings, with the aim of improving the clinical treatment outcomes for patients with gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood this study and voluntarily signed the informed consent form;
2. Be at least 18 years old, regardless of gender;
3. Have histologically and/or cytologically confirmed metastatic or locally advanced gastric or gastroesophageal junction adenocarcinoma, and have experienced at least one failure of systemic treatment (Note: The previously accepted systemic treatment regimens in this protocol include chemotherapy alone or in combination with multiple drugs, or immunotherapy combined with chemotherapy, or failure after receiving anti-HER-2 targeted therapy for HER-2 positive cases. Failure is defined as intolerable toxic side effects, disease progression during treatment, or recurrence after the end of treatment);
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
5. Have an expected survival of ≥ 12 weeks;
6. Have at least one measurable lesion (according to RECIST 1.1);
7. Have normal major organ functions, meeting the following criteria:

1.Blood routine examination: Hemoglobin (Hb) ≥ 90g/L; Absolute neutrophil count (ANC) ≥ 1.5×10⁹/L; Platelet count (PLT) ≥ 100×10⁹/L; White blood cell count (WBC) ≥ 3.0×10⁹/L; 2.Biochemical examination: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5× the upper limit of normal (ULN) (for patients with liver metastasis, ≤ 5×ULN); Serum total bilirubin (TBIL) ≤ 1.5×ULN (for subjects with Gilbert's syndrome, ≤ 3×ULN; for patients with liver metastasis, total bilirubin ≤ 3×ULN); Serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance rate ≥ 50ml/min; 3.Coagulation function: Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN; 4.Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥ 50%; 8.For subjects with potential fertility, they need to use at least one medically approved contraceptive measure (such as an intrauterine device, contraceptive pills, or condoms) during the study treatment period and within 180 days after the end of the study treatment; and the serum/urine human chorionic gonadotropin (HCG) test must be negative before the first administration; and they must not be lactating.

Exclusion Criteria:

1. Have previously received treatment with VEGF or VEGFR inhibitors;
2. Have received live vaccines within 4 weeks before enrollment or are likely to receive them during the study period;
3. Have had an autoimmune disease or a history of autoimmune disease within 4 weeks before enrollment;
4. Have previously received allogeneic bone marrow transplantation or organ transplantation;
5. Have had another malignant tumor within 5 years before enrollment, except for skin basal cell carcinoma or squamous cell carcinoma after radical resection, or cervical carcinoma in situ;
6. Have symptomatic or active central nervous system (CNS) metastases or carcinomatous meningitis (patients with asymptomatic or stable brain metastases after treatment are allowed to be included);
7. Have a history of severe cardiovascular and cerebrovascular diseases:

   * Have experienced cerebrovascular accident (excluding lacunar infarction, mild cerebral ischemia or transient ischemic attack, etc.) within 6 months before the first administration of the study drug, myocardial infarction, unstable angina pectoris, uncontrolled arrhythmia (including QTc interval ≥ 450ms for men and ≥ 470 ms for women) (QTc interval is calculated using the Fridericia formula);
   * Have a New York Heart Association (NYHA) cardiac function classification > grade II or a left ventricular ejection fraction (LVEF) < 50%;
8. Have clinically uncontrolled active infections, such as acute pneumonia, active hepatitis B or hepatitis C (for a history of hepatitis B virus infection, regardless of drug control, hepatitis B virus DNA ≥ 1×10⁴ copies/mL or > 2000 IU/ml);
9. Have uncontrollable malignant ascites (defined as ascites that cannot be controlled by diuretics or puncture as judged by the researcher);
10. Have uncontrolled hypertension that cannot be controlled by drugs currently, defined as systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg (except for patients whose blood pressure can be controlled by dual-drug antihypertensive treatment before enrollment);
11. Have urine routine indicating proteinuria ≥ 2+ and 24-hour urinary protein quantification > 1.0g;
12. Have active ulcers in the stomach and duodenum, digestive tract diseases such as ulcerative colitis, or active bleeding in unresected tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by the researcher;
13. Have active bleeding or a bleeding tendency;
14. Have diseases or conditions that affect the absorption of the drug currently, or be unable to take fruquintinib orally;
15. Have experienced allergic reactions to fruquintinib and/or the excipients in the test drug;
16. Be considered by the researcher as unsuitable for enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 weeks